CLINICAL TRIAL: NCT01795755
Title: The Impact of Horse Assisted Therapy (HAT) on Treatment Outcomes
Brief Title: YATEP - The Impact of Horse Assisted Therapy (HAT) on Treatment Outcomes
Acronym: HAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Swedish-Norwegian Foundation for Equine Research (Unknown); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Espen Walderhaug, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAT-11-1
Record Dates: First submitted 2012-07-06; First posted 2013-02-21 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Addiction
Keywords: Horse Assisted Therapy (HAT); Equine Assisted Psychotherapy (EAP); clinical trial; Randomised Controlled Trial (RCT); psychotherapy
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treat as usual + Horse assisted therapy ( HAT) (Experimental): Treatment as usual means mentalization based inpatient treatment. Horse assisted therapy(HAT) is a structured program of 12 X 90 minute sessions (horse care, ground and mounted work) conducted by two clinically qualified therapists.
  Interventions: Behavioral: Mentalization based inpatient treatment.; Behavioral: Horse assisted Therapy (HAT)
- Treatment as usual (Active Comparator): Treatment as usual means mentalization based inpatient treatment.
  Interventions: Behavioral: Mentalization based inpatient treatment.

INTERVENTIONS:
Behavioral: Mentalization based inpatient treatment. — 1-3 month of inpatient treatment
Behavioral: Horse assisted Therapy (HAT) — A structured program of 12 X 90 minute HAT sessions (horse care, ground and mounted work) conducted by two clinically qualified therapists who are also Level I Riding Instructors.
  Arms: Treat as usual + Horse assisted therapy ( HAT)

SUMMARY:
The objective of the study is to assess the impact of horse assisted therapy (HAT) on:

* Addiction treatment outcomes (its effectiveness as an alternative therapy)
* Addiction treatment dropout & addiction relapse (its efficacy in preventing dropout).

Hypothesis: HAT will correlate with:

* beneficial treatment outcomes of depression, anxiety, aggression
* with improved self esteem & motivation
* lower treatment dropout & addiction relapse.

DETAILED DESCRIPTION:
Background Inclusion of horses in therapeutic settings is a scientific issue with significant social and health implications in Norway. Challenges include increasing provision of horse assisted therapy of variable quality to vulnerable population groups with little substantiating evidence of associated benefit(s) due to lack of research, design issues, mainstream clinicians'/scientists' scepticism of "alternative therapy" and associated difficulties in attracting top researchers and funding. Extensive review of literature found a growing volume of studies but as indicated in the most recent systematic review, there are few studies with adequate research design.

Oslo University Hospital's Dept of Addiction Treatment - Youth (AUA) presents a unique research/evaluation potential to study HAT. It will treat approximately 100 patients per year aged 16 to 26 years with a primary diagnosis of addiction. Horse assisted therapy (using AUA's residential herd) is an integral part of the addiction therapeutic program. Furthermore, AUA's strong emphasis on research and its Youth Addiction Treatment Evaluation Project (YATEP) data base will provide an evidence base needed for sound study in an emerging area of science and psychotherapy.

Patient drop out from addiction therapy is high, often exceeding 50% (Stark 1992). Many AUA patients claim that they remain in treatment because of the horses.

The study is a randomised controlled trial of in-patients undergoing treatment. The Participant Group has treatment as usual plus HAT; the Control Group treatment as usual.

Participant and control groups are drawn from AUA patients (aged 16 to 26 years of age with a primary diagnosis of addiction International Classification of Diseases (ICD F10-F19), admitted between 2013 and 2014 to AUA's in-patient unit and who have consented to participate in research.

HAT is a structured program of 12 X 90 minute therapeutic sessions with horses, including horse care, ground and mounted work, conducted by two clinically qualified therapists who are also Level I Riding Instructors.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of addictionInternational Classification of Diseases ICD F10-F19, admitted in 2011-2014 for treatment at AUA's in-patient unit

Exclusion Criteria:

* Ongoing psychoses

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Lower treatment dropout | Within treatment period of upto 3 months
  Reason for treatment exit, including drop out, is obtained from data recorded in the Department's YATEP data base.

SECONDARY OUTCOMES:
Lower emotional distress (composite measure) | Within the treatment period of upto 3 months
  The measure tests whether depression, anxiety and depression improve with horse assisted therapy (as claimed in non-scientific/popular horse literature). Measurements are taken using Hopkins Symptom Check List (HSCL-25) and Severity Indices of Personality Problems (SIPP-118) from data recorded in the Department's YATEP data base.
Improved self-esteem | Winthin the treatment period of upto 3 months
  The measure tests whether self-esteem improves with horse assisted therapy (as claimed in non-scientific/popular horse literature). Improvement will be measured using the Rosenberg Self Esteem Scale from data recorded in the Department's YATEP data base.

CONTACTS AND LOCATIONS:
Overall Officials: Espen KA Arnevik, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Department of addiction treatment - youth, Oslo, Norway

REFERENCES:
- [Derived] Gatti F, Walderhaug E, Kern-Godal A, Lysell J, Arnevik EA. Complementary horse-assisted therapy for substance use disorders: a randomized controlled trial. Addict Sci Clin Pract. 2020 Feb 4;15(1):7. doi: 10.1186/s13722-020-0183-z. PMID 32019584